CLINICAL TRIAL: NCT01809756
Title: The Effect of Caphosol® on the Development of Esophagitis in (N)SCLC Patients Treated With Concurrent Chemo/Radiotherapy A Prospective Study of Caphosol + Standard of Care Versus Standard of Care
Brief Title: The Effect of Caphosol® on the Development of Esophagitis in (N)SCLC Patients Treated With Concurrent Chemo/Radiotherapy
Acronym: CARACTER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: bad taste of Caphosol - early stop of intake by patients
Sponsor: Amphia Hospital (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, drs. Nils E van 't Veer, ziekenhuisapotheker, drs. (ziekenhuisapotheker), Amphia Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL41938.015.12
Record Dates: First submitted 2013-03-04; First posted 2013-03-13 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Small Cell Lung Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caphosol (Active Comparator)
  Interventions: Other: Caphosol
- No intervention (No Intervention)

INTERVENTIONS:
Other: Caphosol — Caphosol 4 times a day
  Arms: Caphosol

SUMMARY:
Rationale: In the Netherlands 1770 people are being diagnosed with SCLC (Small Cell Lung Cancer) and 8764 patients are being diagnosed with NSCLC (Non Small Cell Lung Cancer) in 2011. This is approximately 15% and 75% of all new diagnosed lungcancers. Part of them will need a combination of chemo-radiationtherapy. A review of the incidence and severity of esophagitis in (N)SCLC patients receiving a combination of chemotherapy and once daily radiotherapy revealed overall esophagitis rates up to 58% experiencing esophagitis grade 2 and higher. As concurrent radiotherapy is moving to twice daily radiation (30 x 1,5 Gy in 3 weeks or 30-35 x 2 Gy in 3 weeks) it is expected that the incidence of esophagitis will rise, the clinical symptoms are likely to arise earlier and become more severe.

Mucositis of the upper tractus digestivus is a serious adverse event leading to pain, problems with swallowing and decreased food intake. It has a negative infect on QoL and can lead to prolonged hospital stay and delayed cancer treatment. Physicians seek improvements in treatment modalities to improve these daily patient toxicities.

Caphosol® is an advanced electrolyte solution indicated as an adjunct to standard oral care in treating oral mucositis caused by radiation or high dose chemotherapy. Positive effects of Caphosol® oral rinse 4 times daily in a study with head and neck chemoradiation patients were found on the presence of mucositis and on oral comfort.

It's supposed that the pathogenesis of chemo- or radiotherapy induced mucositis is the same for the whole tractus digestivus. The appearance does differ due to differences in cell proliferation.

Swallowing Caphosol® after oral rinse could have a positive effect on esophageal mucositis on time of onset, severity and duration.

Objective: Adding the use of Caphosol® (rinsing and swallowing four times a day) to the standard of care for esophagitis/mucositis, reduces the incidence, onset, duration and severity of esophagitis in (N)SCLC patients, comparing to the standard of care alone.

Study design: A multi-centre, open, randomized prospective phase II study. Study population: 108 patients 18 years or older with histologically proven (N)SCLC (all histological subtypes), treated with concurrent chemo- and radiotherapy are estimated to be included in this study (2:1 ratio inclusion; 72 patients with Caphosol® and 36 patients without Caphosol®; α=0.05, power 80%).

Intervention (if applicable): 108 patients eligible for this study will be monitored during their (N)SCLC chemo/radiotherapy treatment. One group of 72 patients will receive Caphosol®, 4 times a day - next to the standard of care. Caphosol® will start at day 1 of treatment and will be continued until 3 weeks after the last radiotherapy (RT).Another group of 36 patients will receive only the current standard of care for esophagitis. The patients will be randomly assigned to one of the groups.

Main study parameters/endpoints: The primary objective is to estimate the incidence, onset, duration and severity of esophagitis in (N)SCLC patients undergoing radiation therapy with chemotherapy who receive Caphosol®.

Secondary study parameters/outcome of the study (if applicable):

1. To correlate components of esophagitis data with clinical outcomes (pain, dysphagia, analgetic use, oral intake, weight loss, infection, need for hospitalization, QoL)
2. Discontinuation or delay of chemotherapy due to esophagitis. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks are very small. The patient has to fill in a Esophagitis Daily Questionnaire and during regular visits QOL questionaires are performed.

Sputumswabs are collected on a weekly basis for determination of the microbiological flora of the mouth. During regular blood control max. 8 ml extra blood is taken for immunologic status research.

Caphosol® is a saturated calciumphosphate solution. The daily intake of calcium and phosphor when swallowing Caphosol® 4 times daily is far beyond the Acceptable Daily Intake (ADI)(< 5%). Compared to daily nutrients like milk (270 mg calcium per unit milk (225 ml)) or meat (200 mg phosphor per 100 g meat) the intake of calcium and phosphor due to Caphosol® is negligible and is considered safe.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients with histologically proven (N)SCLC (all histological subtypes), treated with concurrent chemo- and radiotherapy.
* Ability to understand the protocol and willing to provide written informed consent

Exclusion Criteria:

* Concurrent participation in a clinical trial in which the subject is taking or receiving any investigational agent that may affect the frequency, severity or duration of mucositis.
* Pre-existent esophagitis.
* Receiving investigational treatment for the prevention or treatment of mucositis.
* Prior irradiation to the lung or head and neck region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
number of patients with esophagitis | 3 months after the end of the Caphosolintervention
duration until onset of esophagitis (days) | 3 months after the end of the Caphosolintervention
duration of the period of esophagitis (days) | 3 months after the end of the Caphosolintervention
severity of esophagitis (NCI Common Terminology Criteria for Adverse Events (CTCAE) 4.0 score) | 3 months after the end of the Caphosolintervention

SECONDARY OUTCOMES:
Number of patients who discontinue chemotherapy due to esophagitis. | 3 months after Caphosolintervention
Number of patients with delayed chemotherapy due to esophagitis. | 3 months after Caphosolintervention
QoL (EORTC Quality of Life Questionnaire (QLQ) QLQ-C30 and EORTC QLQ-OES18) | 3 months after Caphosolintervention
dysphagia(NCI CTCAE 4.0 score) | 3 months after Caphosolintervention
analgetic use(NCI CTCAE 4.0 score) | 3 months after Caphosolintervention
oral intake (NCI CTCAE 4.0 score) | 3 months after Caphosolintervention
weight loss (NCI CTCAE 4.0 score) | 3 months after Caphosolintervention

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amphia Hospital, Breda, North Brabant
  - Erasmus Medical Centre, Rotterdam